CLINICAL TRIAL: NCT06656091
Title: Simmitinib Versus Investigator's Choice of Chemotherapy for Participants With Advanced or Metastatic Oesophageal Squamous Cell Carcinoma : a Randomised, Open-label, Multicentre, Phase 3 Study
Brief Title: A Study of Simmitinib Versus Chemotherapy for Participants With Advanced Oesophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1818-008
Record Dates: First submitted 2024-10-14; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Advanced Oesophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: simmitinib 6mg,QD ,3 weeks on 1 week off Control Group：investigator's choice of chemotherapy,include docetaxel or irinotecan.
  docetaxel injection 75mg/m^2,d1,every 3 weeks； ilinotecan injection 180mg/m^2,d1,every 2 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simmitinib (Experimental): simmitinib 6mg,QD ,3 weeks on 1 week off
  Interventions: Drug: simmitinib
- investigator's choice of chemotherapy (Active Comparator): docetaxel injection 75mg/m^2,d1,every 3 weeks；or ilinotecan injection 180mg/m^2,d1,every 2 weeks
  Interventions: Drug: investigator's choice of chemotherapy,include docetaxel or irinotecan.

INTERVENTIONS:
Drug: simmitinib — simmitinib 6mg,QD ,3 weeks on 1 week off
  Arms: simmitinib
Drug: investigator's choice of chemotherapy,include docetaxel or irinotecan. — docetaxel injection 75mg/m^2,d1,every 3 weeks or ilinotecan injection 180mg/m^2,d1,every 2 weeks
  Arms: investigator's choice of chemotherapy

SUMMARY:
To evaluate the overall survival of simmitinib versus investigator's choice of chemotherapy for Participants with advanced or metastatic oesophageal squamous cell carcinoma who have disease progression after first-line standard therapy.

DETAILED DESCRIPTION:
This is a randomised, open-label, multicentre, phase 3 study. Participants with advanced or metastatic oesophageal squamous cell carcinoma who have disease progression after first-line standard therapy will be randomly assigned to the experimental group or control group in a 1:1 ratio. The experimental group received treatment with Simmitinib, while the control group received investigator's choice of chemotherapy, include docetaxel or irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have fully understood and voluntarily sign the ICF for this study; 2. Age of 18-75 years (inclusive), male or female； 3. Histologically or cytologically confirmed esophageal squamous cell carcinoma with locally advanced unresectable, local recurrence or with distant metastasis； 4. Second-line patients with disease progression after only first-line standard therapy（Standard treatment: Chemotherapy with platinum, paclitaxel, or fluorouracil combined with immunosuppressive regimen. Progression during maintenance therapy will be allowed.Concurrent chemoradiotherapy with recurrence or metastasis after surgery is considered as first-line treatment. Progression during Concurrent chemoradiotherapy/ adjuvant/neoadjuvant therapy or within 6 months of the last dose is considered a first-line standard treatment failure）; 5. At least one evaluable lesion according to RECIST 1.1; 6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1; 7. Expected survival is more than 3 months； 8. Have recovered from any prior adverse effects of chemotherapy, surgery, radiation, or other antitumor therapy to CTCAE V5.0 criteria ≤ Grade 1 or baseline (except for toxicity such as hair loss that the investigator determines is not a safety risk)； 9. Adequate organ function, defined as:

  1. Absolute Neutrophil count (ANC) ≥ 1.5 × 10^9/L;
  2. Platelet count (PLT) ≥ 100× 10^9/L;
  3. Hemoglobin (Hb) ≥ 90 g/L;
  4. Serum creatinine ≤ 1.5 × ULN and Creatinine clearance (CCr)≥60mL/min(According to the Cockcroft-Gault formula);
  5. Serum total bilirubin (TBIL) ≤ 1.5 × ULN;
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (≤ 5.0 × ULN for patients with liver metastases);
  7. Prothrombin time (PT)、activated partial thromboplastin time (APTT)、international normalized ratio(INR)≤1.5 × ULN(No previous anticoagulant therapy) 10. Male and female patients of childbearing age must agree to take effective contraceptive measures during treatment and within 6 months after the last dose of treatment. Female participants must have a negative serum or urine pregnancy test result within 7 days prior to randomization and must be non-lactating.

Exclusion Criteria:

* 1. Patients who have previously received any anti-tumor therapy within 4 weeks prior to randomization; 2. Patients who have previously received major surgical treatment、open biopsy、other clinical trial drug treatment or any live attenuated vaccine within 4 weeks prior to randomization, or are expected to received any live attenuated vaccine during the study.

  3. Patients who have previous treatment with anti-angiogenic drugs (such as anlotinib, apatinib, Fruquintinib, Surufatinib, Bevacizumab, etc.) 4. LVEF <50%； 5. BMI≤18.5 kg/m^2； 6. Symptomatic central nervous system (CNS) metastases or meningeal metastases 7. Patients with other types of malignant tumors within 5 years prior to the screening, except for radically resected, non-recurrent skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ, or other carcinoma in situ； 8. Patients with bleeding tendency; active bleeding or a history of heavy bleeding within the past 6 months； 9. Urine protein ≥ ++ and 24 h urine protein > 1.0 g at screening period； 10. Presence of any severe and/or uncontrolled disease before starting treatment； 11. Patients with Liver cirrhosis or active hepatitis； 12. Patients with abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or abdominal abscess within 6 months before randomization； 13. Patient previously had or currently has a mental disorder or suffers from epilepsy and requires treatment； 14. Patients had prior retinal pigment epithelial detachment or have evidence of ongoing retinal pigment epithelial detachment； 15. Any active infection requiring antibiotics or hormones systemic treatment by intravenous infusion within 14 days prior to randomization; 16. Patients had prior interstitial lung disease,or have evidence of active non-infectious pneumonia treated with corticosteroids； 17. Inability to swallow drugs orally, or presence of clinically significant gastrointestinal disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
OS | up to approximately 3 years

SECONDARY OUTCOMES:
ORR | up to approximately 3 years
  Objective Response Rate (ORR) evaluated by investigators based on RECIST 1.1
PFS | up to approximately 3 years
  Progression-free Survival
DCR | up to approximately 3 years
  Disease Control Rate
DOR | up to approximately 3 years
  Duration of Objective Response
AE | From first dose to 28 days post the last dose
  Incidence rate of Adverse Event
FGF19 protein expression, FGF gene amplification status | baseline
  IHC detection of FGF19 protein expression in tumor tissues FISH detection of FGF19 gene amplification status in tumor tissues NGS detection of FGF-FGFR pathway related gene status, including gene amplification, mutation, or fusion
PK | Cycle 1 Day 1 to Cycle 2 Day 15 (each cycle is 28 days)
  Plasma Concentration of simmitinib

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No